CLINICAL TRIAL: NCT05009173
Title: LiPSTICk Trial-Lumbar Puncture Stylet Technique in Children; A Randomized-controlled Study
Brief Title: Lumbar Puncture Stylet Technique in Children
Acronym: LiPSTICk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Ariane Boutin MD, MSc FRCPC, Principal investigator, St. Justine's Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: Stylet in:out
Record Dates: First submitted 2021-03-17; First posted 2021-08-17 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Traumatic Tap
Keywords: Lumbar puncture; Stylet-in; Stylet-out; Children; Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stylet-in (Active Comparator): Lumbar puncture performed keeping the stylet inside the needle until the practitioner reaches the appropriate location.
  Interventions: Procedure: Lumbar puncture using the stylet-in technique
- Stylet-out (Active Comparator): The practitioner remove the stylet once he/she has passed the skin and moves the needle forward with the stylet.
  Interventions: Procedure: Lumbar puncture using the stylet-out technique

INTERVENTIONS:
Procedure: Lumbar puncture using the stylet-in technique — This method consists of inserting the needle with the stylet-in, then only remove the stylet once the desired depth is achieved and CSF flow is expected. If no CSF comes back, the stylet is replaced before continuing to advance the needle until the subarachnoid space is entered. This is the technique generally used in our emergency department and will serve as the control treatment group.
  Arms: Stylet-in
Procedure: Lumbar puncture using the stylet-out technique — This method consists of inserting the needle through the epidermis and the dermis, which is estimated as a 0.5 to 1 cm length in children, then remove the stylet before progressing through the other structures until the subarachnoid space is entered. This approach will be used in the experimental technique group.
  Other Names: Lumbar puncture using the early stylet removal technique
  Arms: Stylet-out

SUMMARY:
Lumbar puncture (LP) is a procedure performed frequently among children in the emergency department (ED). Although it has been performed for decades, and for distinct indications, the technique itself can often lead to traumatic results, which can complicate its interpretation and lead to over-treatments and hospitalizations. Several factors have been suggested to improve the success rate of LPs. Among them, the stylet-out (SO), also known as the early stylet removal technique, has been suggested but not properly studied.

The aim of this study is to evaluate whether the stylet-out technique can reduce the probability of failure or traumatic lumbar puncture procedures in a pediatric population presenting to the emergency department as compared to the standard stylet-in (SI) approach.

To achieve this goal, the investigator will conduct a randomized controlled trial comparing the SO versus SI techniques in a tertiary care, pediatric, university-affiliated emergency. All children younger than 18 years of age requiring a LP as part of their ED workup will be eligible and randomized to either the standard SI or SO group. The primary outcome will be the first-attempt LP success rate as defined by the minimum amount of cerebrospinal fluid (CSF) necessary to perform a leukocyte count and bacterial/viral CSF cultures, according to each laboratory with red blood cell count < 1000/mm3. Secondary outcomes will include the following: overall LP success rate (i.e. despite number of attempts), proportion of traumatic LP, number of LP attempts, number of changes in providers performing the LP, proportion of traumatic LP, total time to procedure, mean difference in pain scores and satisfaction rates in both groups.

The hypothesis is that the use of the Stylet Out approach will reduce the number of failed and traumatic LP in the pediatric population presenting to the ED as compared to the standard SI approach.

ELIGIBILITY:
Inclusion Criteria:

* All patients younger than 18 years of age (no minimal age)
* All patients who require a diagnostic lumbar puncture as part of their emergency department workup

Exclusion Criteria:

* Patients with lumbar puncture contraindications
* Parents/patients unable to give consent
* Patients who have had a traumatic of failed lumbar puncture prior to the emergency department transfer

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 395 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
First-time lumbar puncture success rate | 1 hour after procedure
  Defined as the minimum amount of CSF necessary to perform a leukocyte count and a CSF bacterial/viral culture, according to the hospital laboratory, with a red blood cell count <1,000/mm3

SECONDARY OUTCOMES:
Lumbar puncture success rate despite the number of attempts | 1 hour after procedure
  Defined as the minimum amount of CSF necessary to perform a leukocyte count and CSF bacterial/viral culture according to each laboratory with red blood cell count <1,000/mm3
Proportion of final traumatic lumbar puncture | 1 hour after procedure
  Defined as a red blood cell count > 1,000/mm3 not explained by a concomitant meningitis diagnosis (i.e. negative culture)
Number of lumbar puncture attempts in total | immediately after procedure
  Defined as any time a needle that is completely outside the body penetrates the skin
Number of changes in provider performing the lumbar puncture | immediately after procedure
  The first provider could be a trainee, and then a trained physician
Length of procedure | immediately after procedure
  Measured from the time the needle pierces the skin until first drop of CSF
Mean difference in Evendol pain scores and NRS-11 scores | during procedure
  Evendol pain scores will be applied for all patients and NRS-11 will be applied for children 6 years and older remembering the procedure
Satisfaction with procedure | immediately after procedure
  LP provider satisfaction as measured by a five-point Likert Scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No